CLINICAL TRIAL: NCT07308704
Title: DELINEATE-Deploy: Deep Learning for Echo Analysis, Tracking, and Evaluation - Prospective Deployment Platform IRB
Brief Title: A Study Of Deep Learning For Echo Analysis, Tracking, And Evaluation
Status: Not yet recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tim Poterucha, Principal Invetigator, Mayo Clinic
Other Study IDs: 25-007929
Record Dates: First submitted 2025-12-17; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cardiomyopathy; Ischemic Heart Disease; Cardiac Amyloidosis
MeSH Terms: conditions — Cardiomyopathies; Myocardial Ischemia; Amyloid Neuropathies, Familial | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Genetic cardiomyopathy arm
  Interventions: Diagnostic Test: Transthoracic Echocardiography (TTE)
- Ischemic cardiomyopathy arm
  Interventions: Diagnostic Test: Transthoracic Echocardiography (TTE)
- Cardiac amyloidosis arm
  Interventions: Diagnostic Test: Transthoracic Echocardiography (TTE)
- Hypertrophic cardiomyopathy (HCM) arm
  Interventions: Diagnostic Test: Transthoracic Echocardiography (TTE)

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiography (TTE) — AI analysis of transthoracic echocardiography to improve disease detection.

SUMMARY:
The purpose of this study is to deploy and evaluate informational AI-Echo algorithms that assist echo clinicians in interpreting core echocardiographic parameters (e.g., LV/RV size and function, valvular disease severity) and stratifying disease progression risk. The primary outcome is clinician usability, interpretive consistency, and workflow integration. Second, we will conduct a pragmatic, stepped-wedge clinical trial with multiple arms evaluating diagnostic AI-Echo algorithms designed to identify specific cardiovascular diseases- such as genetic cardiomyopathy, ischemic heart disease, and cardiac amyloidosis-and assess whether AI deployment increases diagnostic testing and shortens time to diagnosis. Trials will be conducted using EHR-based notification systems with cluster-level randomization.

ELIGIBILITY:
Inclusion criteria:

* Genetic cardiomyopathy arm: Clinicians who order, perform, and interpret echocardiograms and act on echocardiogram results, including both physicians and allied health staff taking care of patients aged ≥18 years who are undergoing a comprehensive TTE at a participating Mayo Clinic site with AI-Echo analysis indicating high risk for a genetic cardiomyopathy. A high-risk score will be defined by a specific threshold determined in model development to maximize sensitivity while maintaining an adequate positive predictive value to support clinical deployment
* Ischemic cardiomyopathy arm: Clinicians who order, perform, and interpret echocardiograms and act on echocardiogram results, including both physicians and allied health staff taking care of patients aged ≥18 years who are undergoing a comprehensive TTE with AI-Echo analysis indicating high risk for ischemic cardiomyopathy. A high-risk score will be defined by a specific threshold determined in model development to maximize sensitivity while maintaining an adequate positive predictive value to support clinical deployment.
* Cardiac amyloidosis arm: Clinicians who order, perform, and interpret echocardiograms and act on echocardiogram results, including both physicians and allied health staff taking care of patients aged ≥18 years who are undergoing a comprehensive TTE with AI-Echo analysis indicating high risk for cardiac amyloidosis. A high-risk score will be defined by a specific threshold determined in model development to maximize sensitivity while maintaining an adequate positive predictive value to support clinical deployment.
* Hypertrophic cardiomyopathy (HCM) arm: Clinicians who order, perform, and interpret echocardiograms and act on echocardiogram results, including both physicians and allied health staff caring for patients aged ≥18 years who are undergoing a comprehensive TTE at a participating Mayo Clinic site, with AI-Echo analysis indicating high risk for HCM. A high-risk score will be defined by a specific threshold determined during model development to maximize sensitivity while maintaining adequate positive predictive value for clinical deployment.

Exclusion criteria:

* Genetic cardiomyopathy arm: Studies performed within the past 2 years at a Mayo site or in those patients with known or suspected diagnosis of genetic cardiomyopathy under evaluation, on hospice care, or who have an expected non-cardiac life expectancy <1 year, and patients who have opted out of institutional and state research authorizations.
* Ischemic cardiomyopathy arm: Studies performed within the past 2 years at a Mayo site or in those patients with known CAD; prior myocardial infarction; revascularization with PCI or CABG; ischemic testing within the past 12 months; hospice care or expected non-cardiac life expectancy <1 year, and patients who have opted out of institutional and state research authorizations.
* Cardiac amyloidosis arm: Studies performed within the past 2 years at a Mayo site or in those patients with prior amyloid-specific testing (e.g., technetium pyrophosphate scan, cardiac MRI with late gadolinium enhancement suggestive of amyloid) or biopsy-proven systemic amyloidosis, on hospice care, or have expected non-cardiac life expectancy <1 year, and patients who have opted out of institutional and state research authorizations.
* Hypertrophic cardiomyopathy (HCM) arm: Studies performed within the past 2 years at a Mayo site or patients with a known diagnosis of HCM documented in the medical record prior to the index TTE, prior septal reduction therapy (surgical myectomy or alcohol septal ablation), or patients on hospice care or with an expected non-cardiac life expectancy <1 year, and patients who have opted out of institutional and state research authorizations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinicians who order, perform, and interpret echocardiograms and act on echocardiogram results, including both physicians and allied health staff taking care of patients aged ≥18 years.
Sampling Method: Non-Probability Sample
Enrollment: 10040000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients diagnosed with genetic cardiomyopathy confirmed by genetic testing | Baseline
  Number of patients in the genetic cardiomyopathy arm who have a confirmed diagnosis of genetic cardiomyopathy based on genetic testing. Confirmation requires identification of a pathogenic or likely pathogenic variant in a cardiomyopathy-associated gene.
Number of patients diagnosed with obstructive coronary artery disease | Baseline
  Number of patients diagnosed with obstructive coronary artery disease in the ischemic cardiomyopathy arm, defined as ≥70% stenosis in any epicardial vessel, ≥50% in the left main coronary artery on coronary CTA or invasive angiography, or evidence of ≥3 ischemic myocardial segments on stress testing or high-risk perfusion features such as transient ischemic dilation.
Number of patients diagnosed with cardiac amyloidosis | Baseline
  Number of patients diagnosed with cardiac amyloidosis in the cardiac amyloidosis arm confirmed by consensus criteria, both imaging- and pathology-based amyloidosis diagnostic pathways.
Number of patients diagnosed with hypertrophic cardiomyopathy | Baseline
  Number of patients diagnosed with hypertrophic cardiomyopathy in the hypertrophic cardiomyopathy (HCM) arm according to standard guideline-based criteria (e.g., unexplained LV wall thickness ≥15 mm, or ≥13 mm in first-degree relatives, in the absence of other causes of hypertrophy).

SECONDARY OUTCOMES:
Time from index TTE to confirmed diagnosis | Baseline
  Time from index TTE to confirmed diagnosis of hypertrophic cardiomyopathy, cardiac amyloidosis, obstructive coronary artery disease, or genetic cardiomyopathy. Measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Poterucha, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No